CLINICAL TRIAL: NCT00601653
Title: CBT and Dieting: Effects on Psychopathology and Weight in BED
Brief Title: Effectiveness of Cognitive Behavioral Therapy Plus Nutritional Counseling in Promoting Weight Loss in People With Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0706002747; 5R21MH082629 (NIH); DATR A2-AID
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Binge Eating Disorder; Obesity; Overweight
Keywords: Binge Eating Disorder; BED; Nutrition; Energy Density; Cognitive Behavioral Therapy; CBT
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Overweight | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cognitive behavioral therapy plus general nutrition counseling
  Interventions: Behavioral: Cognitive behavioral therapy plus general nutrition counseling (CBT+GN)
- 2 (Experimental): Cognitive behavioral therapy plus low energy density diet counseling
  Interventions: Behavioral: Cognitive behavioral therapy plus low energy density diet counseling (CBT+LED)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy plus general nutrition counseling (CBT+GN) — CBT+GN includes 21 sessions over 6 months. Each treatment session includes 40 minutes of CBT and 20 minutes of nutritional counseling.
  Arms: 1
Behavioral: Cognitive behavioral therapy plus low energy density diet counseling (CBT+LED) — CBT+LED includes 21 sessions over 6 months. Each treatment session includes 40 minutes of CBT and 20 minutes of nutritional counseling that centers upon eating higher volumes of low-calorie foods.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of adding nutritional counseling to cognitive behavioral therapy in treating obese people with binge eating disorder.

DETAILED DESCRIPTION:
Binge eating disorder (BED) is one of the most common eating disorders, with millions of affected Americans. The majority of people who binge eat are mildly to severely overweight, but people of normal weight can also have BED. People with BED frequently eat excessive amounts of food in a short period of time, often feeling a loss of control over their urge to eat. Following a binge eating episode, the person usually experiences feelings of guilt, depression, embarrassment, and disgust. Beyond the psychological distress caused by binge eating, people who binge eat are at a higher risk for more serious health problems associated with weight gain, including high blood pressure, diabetes, heart disease, high cholesterol, and stroke. Previous studies on BED have found cognitive behavioral therapy (CBT) to be the most effective treatment in improving binge eating habits, attitudinal features of eating disorders, and psychological functioning. However, CBT alone has not been nearly as effective in producing clinically significant weight loss in those who are overweight. This study will evaluate the effectiveness of adding nutritional counseling to CBT in treating obese people with BED.

Participants in this 1-year study will be randomly assigned to one of two treatment groups: CBT plus general nutrition counseling (CBT+GN) or CBT plus low energy density diet counseling (CBT+LED). All participants will receive 21 hourly individual treatment sessions over a 6-month period. Sessions will be weekly for Weeks 1 to 16 and every other week for Weeks 17 to 26. Each treatment session will include 40 minutes of CBT and 20 minutes of nutritional counseling (GN or LED). Assessments will include interviews and questionnaires about symptoms and height and weight measurements. These assessments will occur at baseline, monthly during treatment, and at 6 months post-treatment. At the end of treatment, participants will also have blood drawn to determine lipid levels and will be asked to complete two food intake interviews by phone.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 30
* Meets DSM-IV criteria for BED

Exclusion Criteria:

* Co-existing physical and/or psychiatric conditions that require different treatments than CBT (e.g., bipolar disorder, psychotic illnesses), and/or require more intensive treatment or hospitalization (e.g., suicidality, severe mood disorders)
* Meets criteria for current substance abuse or dependence
* Currently receiving psychiatric, psychological, behavioral, or pharmacologic treatment that is known to affect weight or eating
* Any physical conditions, such as diabetes, known to affect weight or eating
* Pregnant, breastfeeding, or plans to become pregnant during the treatment period
* Cardiac disease, including ischemic heart disease, congestive heart failure, conduction abnormalities, or a history of heart attack
* Serious neurologic illnesses (e.g., seizure history) or medical illnesses (e.g., impaired hepatic or renal function)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | Measured at Year 1

SECONDARY OUTCOMES:
Outcomes related to binge eating disorder (e.g., binge eating, attitudinal features of eating disorders, psychological functioning) | Measured at Year 1
Outcomes related to energy density (e.g., energy density, caloric intake, fat intake, fruit and vegetable consumption, hunger) | Measured at Year 1
Health status (e.g., lipid profile, blood pressure) | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Robin M. Masheb, PhD, Principal Investigator — Yale University

REFERENCES:
- [Result] Masheb RM, Grilo CM, Rolls BJ. A randomized controlled trial for obesity and binge eating disorder: low-energy-density dietary counseling and cognitive-behavioral therapy. Behav Res Ther. 2011 Dec;49(12):821-9. doi: 10.1016/j.brat.2011.09.006. Epub 2011 Sep 28. PMID 22005587